CLINICAL TRIAL: NCT00666640
Title: Parameters Derived From DXA-based Structural Engineering Models of the Proximal Femur as a Biomarker for Hip Fracture Prediction.
Brief Title: 3D Imaging of the Hip Using DXA
Acronym: 3DScans
Status: Completed | Type: Observational
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: Medical Research Council (Other Government); Hologic, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: STH14748
Record Dates: First submitted 2008-04-23; First posted 2008-04-25 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2014-09

CONDITIONS: Osteoporosis; Low-energy Trauma Fracture
Keywords: Osteoporosis; Fracture; DXA; Dual energy x-ray absorptiometry; Computed tomography; 3D DXA
MeSH Terms: conditions — Osteoporosis; Fractures, Bone

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: 50 subjects who have suffered a hip fracture
  Interventions: Device: DXA scan of hip; Device: CT scan of hip
- 2: 50 age matched controls
  Interventions: Device: DXA scan of hip; Device: CT scan of hip

INTERVENTIONS:
Device: DXA scan of hip — Dual-energy X-ray Absorptiometry scan
Device: CT scan of hip — Computed Tomography scan

SUMMARY:
The study aims to determine the efficacy and best methods for predicting hip fractures and diagnosing post-menopausal osteoporosis using three dimensional structural engineering models (SEMs) of proximal femoral bone produced using a Hologic Discovery duel-energy x-ray absorptiometry scanner and Hologic's new 3D Hip(TM) software in comparison to three dimensional SEMs produced using quantitative computed tomography - the current gold standard.

DETAILED DESCRIPTION:
Bone mineral density (BMD) measurements by dual-energy x-ray absorptiometry (DXA) have been available to the clinician for the past 20 years and their use forms the basis of current clinical practice guidelines. The measurements are very useful, but they could be improved upon by taking into account the third dimension of bone (depth) and the distribution of mineral within bone. The value of a diagnostic test depends greatly on the strength of association of the measurement with the outcome. If we find that our new approach strengthens the ability of hip DXA measurements to predict fracture then we will have a greatly improved diagnostic test and so can better identify those patients we should treat. Further, such a test would allow better evaluation of new therapies for osteoporosis, particularly those that may alter bone geometry, including anabolic agents such as teriparatide.

Patients attending for study visits will complete a basic questionnaire to collect information on their bone health and lifestyle (the current Metabolic Bone Centre standard questionnaire). Patients will also undergo DXA scans of their hips on a Hologic Discovery DXA machine using a new 3D imaging technique called '3D HipTM'. Hologic will process 3D HipTM scans and provide us with volumetric dataset of the scans before they provide us with a high performance PC and software for us to do the process on-site. They have already installed the software upgrade and necessary hardware to our Discovery densitometry system to enhance the 3D HipTM capability. Patients will attend for a CT scan of their hip at the medical imaging department of the Northern General Hosptial as per standard practice.

50 postmenopausal women who have recently suffered a hip fracture will be recruited to the study. 50 postmenopausal age matched controls will also be recruited. Subjects will give informed consent and a study visit will be arranged for them to attend for a DXA scan and a CT scan. At the study visit basic demographic data and a brief medical history will be collected on study specific Case Report Forms (CRF).

The intended outcomes of the study are 1) To establish the diagnostic accuracy for hip fracture of the 3D HipTM and SEMs derived from the 3D HipTM, and to determine how much better the 3D HipTM is over the traditional 2D DXA in a case controlled study. 2) To compare three dimensional SEMs of the proximal femur derived from 3D Hip(TM) against simulated SEMs derived using quantitative computed tomography.

ELIGIBILITY:
Inclusion Criteria:

* be female
* at least 5 years post menopausal but <85 years
* be sufficiently mobile to undergo DXA and QCT scanning
* be able and willing to participate in the study and provide written informed consent

Exclusion Criteria:

* bi-lateral hip replacement
* have hip replacement on the non-fractured side
* have any history of cancer within the past 5 years excluding skin cancer non melanomas
* have a history of ongoing conditions or diseases known to cause abnormalities of calcium metabolism or skeletal health (secondary osteoporosis)
* have a history of chronic renal disease (as defined by a creatinine clearance of ≤ 30ml/min)
* Acute or chronic hepatic disease
* Malabsorption syndromes
* Hyperthyroidism as manifested by TSH outside the lower limit of the normal range
* Hyperparathyroidism
* Hypocalcemia or hypercalcemia
* Osteomalacia
* Cushing's syndrome
* patients who are currently on glucocorticoid therapy
* have a history of any known condition that would interfere with the assessment of DXA or CT of hip
* have markedly abnormal clinical laboratory parameters that are assessed as clinically significant by the investigator
* have participated in another clinical trial involving active therapy 3 months prior to randomisation
* have a known confusional state or dementia as documented in hospital notes, or be unsuitable for approach in the opinion of the physician with duty of care

Ages: 50 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community Sample Subjects recruited from A+E attendances/fracture clinics at Sheffield hospitals
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2008-05; Primary Completion 2011-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
To establish the diagnostic accuracy for hip fracture of the 3D HipTM and SEMs derived from the 3D HipTM, and to determine how much better the 3D HipTM is over the traditional 2D DXA in a case controlled study. | 2 years

SECONDARY OUTCOMES:
The secondary outcome measures are parameters related to the hip structure, such as volumetric bone mineral density, cross sectional area, moment of inertia, section modulus, cortical thickness and buckling ratio. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Lang Yang, Dr, Study Director — Sheffield University; Eugene McCloskey, Dr, Study Director — Sheffield University
Locations (1):
- Bone Biomedical Research Unit, Northern General Hospital, Sheffield, South Yorkshire, United Kingdom